CLINICAL TRIAL: NCT03287453
Title: Screen to Save Initiative
Brief Title: Educational Intervention - Improving Knowledge and Screening Rates for Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Electra Paskett, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: OSU-17069; NCI-2017-01357 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2017-09-13; First posted 2017-09-19 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2023-10

CONDITIONS: Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Screening (educational intervention) (Experimental): Participants attend educational sessions comprising of an inflatable colon interactive exhibit that allows visitors to walk through a colon while seeing images, a PowerPoint presentation that contains messages that are tailored to meet the cultural and linguistic needs of Black/African Americans, Appalachians, and Hispanics/Latinos, and or flip books/flip charts. Participants also receive a copy of the study information sheet which contains the basic elements of informed consent and a pre-education session knowledge survey.
  Interventions: Other: Educational Intervention; Other: Survey Administration

INTERVENTIONS:
Other: Educational Intervention — View an inflatable colon interactive exhibit, PowerPoint presentation, flip books, and flipcharts
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial studies how well educational intervention works in improving knowledge and screening rates of colorectal cancer. An educational intervention, such as viewing an inflatable colon, PowerPoint presentation, or flip books/flipcharts, may help improve knowledge about colorectal cancer and how often people get checked for colorectal cancers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To increase colorectal cancer (CRC) knowledge, attitudes, positive behavior change, intent for screening, and screening among at-risk groups.

OUTLINE:

Participants attend educational sessions comprising of an inflatable colon interactive exhibit that allows visitors to walk through a colon while seeing images, or a PowerPoint presentation that contains messages that are tailored to meet the cultural and linguistic needs of Black/African Americans, Appalachians, and Hispanics/Latinos, and flip books/flip charts. Participants also receive a copy of the study information sheet which contains the basic elements of informed consent and a pre-education session knowledge survey.

ELIGIBILITY:
Inclusion Criteria:

* Participants from Franklin County or from Appalachia Ohio (depending on program location)

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2017-04-08 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Change in knowledge and degree to which reported intentions regarding colorectal cancer screening are related to the educational session | Up to two years
  Change in knowledge will be examined as a function of the important covariates: race/ethnicity, sex, age, education and primary language. A paired t-test or Wilcoxon signed-rank test will be used to determine whether there is a statistically significant difference in pre and post session scores. The paired t-test provides a hypothesis test to determine whether pre and post session assessment mean scores differ from each other in a significant way under the assumptions that the paired differences are independent and identically normally distributed. The test statistic is t with n-1 degrees of f
Change in knowledge and strength of intention to be screened | Up to two years
  Will be correlated with key outcomes, specifically actual screening and actions promoting colorectal cancer screening (e.g., encouraging colorectal screening with family/friends). Multivariable logistic regression analyses will be conducted to examine the impact of knowledge change and strength of intentions on these binary outcomes (screened/not screened and encouraged/did not encourage colorectal screening) controlling for important covariates such as sex, race/ethnicity, age, education and primary language. A paired t-test or Wilcoxon signed-rank test will be used to determine whether there
Frequency of reported family history of colorectal cancer | Up to two years
  Will be described in total and as a function of specific racial/ethnic groups.
Participants' plans for future screening | Up to two years
  Will examine relationships between stated plans and key covariates.
Reasons reported for not obtaining colorectal screening | Up to two years
  Response categories will be examined by key covariates.
Self-reported intentions to engage in behavior change to reduce risk of colorectal cancer | Up to two years
  Will be examined by race/ethnicity, sex, education, and health insurance/healthcare coverage.

CONTACTS AND LOCATIONS:
Overall Officials: Electra Paskett, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu